CLINICAL TRIAL: NCT01624298
Title: A Randomized Control Trial to Determine the Effectiveness of Trauma Focused Cognitive Behavioral (TF-CBT) Among Children in Lusaka, Zambia
Brief Title: Randomized Control Trial on Trauma Focused CBT in Zambia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TFCBTRCTDCOF
Record Dates: First submitted 2012-06-18; First posted 2012-06-20 (Estimated); Results first posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-02

CONDITIONS: Post Traumatic Stress Disorder; Depression; Risk Behaviors
Keywords: Randomized controlled trial; Traumatized youth; HIV risk
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Risk-Taking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Wait List Control Group (No Intervention): The wait list control group will be asked to wait for approximately 4 1/2 months before being reassessed and then, unless found to be ineffective or harmful, receive the intervention being provided by the counselor.
- Intervention Group (Experimental): Children randomized into the intervention group will immediately receive the Trauma Focused Cognitive Behavioral Therapy with a trained counselor for 12 weeks.
  Interventions: Behavioral: Trauma Focused Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Trauma Focused Cognitive Behavioral Therapy — TF-CBT (www.musc.edu/tfcbt) is a therapy that helps children/youth ages 5-18 years and their families who have been affected by traumatic events and/or traumatic grief. Components include psychoeducation, relaxation, affective modulation, cognitive processing, Trauma Narrative (gradual exposure), In-vivo exposure, Con-joint session, and Enhancing safety skills. Youth and caregivers are seen once a week for approximately 12 weeks.
  Other Names: TF-CBT
  Arms: Intervention Group

SUMMARY:
The purpose of this study is to study the effectiveness of Trauma Focused Cognitive Behavioral Therapy in subset of children who are affected by trauma with significant mental health symptomatology in order to 1) examine the effectiveness of TF-CBT in reducing the severity of mental health symptoms experienced by traumatized children and adolescents in Lusaka and 2) determine the effectiveness of TF-CBT in reducing HIV risk taking behaviors and increasing coping strategies and health promotion activities in traumatized children and adolescents in Lusaka. The study will be integrated into current programing of the Serenity Harm Reduction Programme, a community and faith based organization focusing on mental health and substance use prevention and treatment, and its partners in 5 compounds.

DETAILED DESCRIPTION:
In preparation for the trial, in February and March of 2012, a US-based clinical psychologist and expert trainer in TF-CBT traveled to Lusaka Zambia and trained 20 counselors in TF-CBT. This included supplemental training of the already established and trained national TF-CBT supervisors from SHARPZ and the University of Zambia (UNZA). Counselors will take on 1 practice case each in TF-CBT. Local supervisors will meet with the counselors in groups on a weekly basis to monitor the intervention and will be in regular phone and email contact to assist with the initiation of cases. The US-based TF-CBT experts (Drs. Murray and Dorsey) will be in contact with the supervisors on a weekly basis (via skype) to assist with the supervision and provide ongoing support to the supervisors and the counselors. This follows the Apprenticeship Model of Training and Supervision (Murray et al., 2011).

As part of the study, 11 assessors will be trained on a comprehensive intake assessment process. The process uses an adapted initial intake form that is currently used by the partner organization to collect basic demographic, health, and other information about the client and a parent or guardian and adds a standard mental health and functioning assessment instrument based on the earlier qualitative and quantitative research conducted by the Johns Hopkins University (JHU) faculty. All children age 5-8 enrolled in the study will receive the demographics section, the PTSD-RI and the Shame measures as well as section one of the World AIDS Foundation measure that covers the topics of HIV Testing and Substance Abuse. Children ages 12 years and older will also receive the World Aids Foundation (WAF) questionnaire section 2 that asks questions related self-efficacy and sexual relationships and violence. Only children ages 12 and older who report yes to having experienced sexual intercourse of any form will be asked section 3 of the WAF which includes questions related to their relationship with their partner, sexual behaviors and HIV-risk behaviors commonly connected to trauma and mental health symptoms. Adults participating in the study will be given a demographics section, a section related to services received and the Child Behavior Checklist (CBCL).

The proposed study will be embedded within the ongoing SHARPZ program. We will study the effectiveness of TF-CBT for children who are affected by trauma with significant mental health symptomatology. The partner organizations will continue to provide services to anyone who seeks their services regardless of whether they meet eligibility for our proposed study, however those who meet our inclusion criteria will be invited to participate in the research component of the SHARPZ service program.

Qualitative exit interviews: Following completion of the therapy by the first set of 20 participants, assessors will ask these intervention participants what has changed since the intervention began and what change they attribute to the intervention. Interviews will be open ended, written by the assessors (not tape recorded) and identifying information will not be recorded. The research team will review these qualitative exit interviews to identify any unexpected positive or negative effects of the intervention. Questions on the more significant and/or frequent responses will be added to the original assessment instrument.

Post-intervention quantitative assessments will be done with the expanded assessment instrument (see qualitative exit interviews above). All post intervention quantitative interviews (including with the wait controls) will be conducted approximately 2-3 weeks after the client has completed the intervention or control period (approximately 12-14 weeks). Those randomized to the intervention will also receive a second post assessment 4 months after receiving the first post assessment. Control cases will only receive one post assessment after the wait list period so that they may then receive the intervention, unless found to be harmful or ineffective, as soon as their wait list period is over.

Following completion of the trial, the data will be analyzed, and if the intervention is found to be effective, it will become a permanent part of the services provided by the counselors at SHARPZ and the partner organizations.

ELIGIBILITY:
Inclusion Criteria:

* Youth found to exhibit significant trauma symptomatology as evidenced by a score of 38 or above on the previously validated PTSD-RI symptom scale (Murray, et al. 2011) (trauma severity is the main study outcome) will be invited to join the trial. Youth must live in Lusaka, Zambia.

Exclusion Criteria:

* Youth currently receiving psychiatric care
* Youth who are actively suicidal
* Persons who are not mentally competent to give assent or whose legal guardians are not mentally competent to give consent to participate in the intervention

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 257 (Actual)
Dates: Start 2012-08; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura K Murray, PhD, Principal Investigator — Johns Hopkins University; Paul Bolton, MBBS MPH, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Serenity Harm Reduction Programme Zambia, Lusaka, Zambia

REFERENCES:
- [Derived] Murray LK, Skavenski S, Kane JC, Mayeya J, Dorsey S, Cohen JA, Michalopoulos LT, Imasiku M, Bolton PA. Effectiveness of Trauma-Focused Cognitive Behavioral Therapy Among Trauma-Affected Children in Lusaka, Zambia: A Randomized Clinical Trial. JAMA Pediatr. 2015 Aug;169(8):761-9. doi: 10.1001/jamapediatrics.2015.0580. PMID 26111066

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began August 15, 2012 and ran until August 1, 2013. Recruitment was done at 5 community organizations located in Lusaka Zambia.
Groups:
- Intervention Group: Children randomized into the intervention group will immediately receive the Trauma Focused Cognitive Behavioral Therapy with a trained counselor for 12 weeks.
  Trauma Focused Cognitive Behavioral Therapy (TF-CBT) is a therapy that helps children/youth ages 5-18 years and their families who have been affected by traumatic events and/or traumatic grief. Components include psychoeducation, relaxation, affective modulation, cognitive processing, Trauma Narrative (gradual exposure), In-vivo exposure, Con-joint session, and Enhancing safety skills. Youth and caregivers are seen once a week for approximately 12 weeks.
Period: Overall Study
Arm/Group | Wait List Control Group | Intervention Group
Started | 126 | 131
Completed | 104 | 106
Not Completed | 22 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Wait List Control Group | Intervention Group | Total
Number analyzed (Participants) | 126 | 131 | 257
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.29 (2.99) | 14.02 (2.78) | 13.66 (2.90)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 121 | 122 | 243
  Between 18 and 65 years | 5 | 9 | 14
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 63 | 128
  Male | 61 | 68 | 129
Region of Enrollment [Number; unit: participants]
  Zambia | 126 | 131 | 257

OUTCOME MEASURES:

1. Primary Outcome: Post Traumatic Stress Disorder- Reaction Index (RI)
Description: The PTSD-RI assesses specific traumatic events a child has experienced or witnessed, and the associated mental health symptoms to such stressors. PTSD-RI can range from a score of 0 on the scale to a score of 4 on the scale. Higher scores are associated with greater symptomatology. The psychometric properties have been extensively demonstrated in the US and Internationally. The PTSD RI has also been translated into three local Zambian languages (Nyanja, Bemba and Tonga) and validated in Zambia in Johns Hopkins University faculty preliminary studies.
Time Frame: Baseline and Follow-up within one month of treatment completion. For controls follow up was 4 months post baseline.
Measure: Mean (Standard Deviation); unit: trauma score
Arm/Group | Wait List Control Group | Intervention Group
Number analyzed (Participants) | 104 | 106
trauma score
  Baseline | 1.75 (0.44) | 1.88 (0.51)
  Post Assessment | 1.38 (0.66) | 0.34 (0.43)

2. Secondary Outcome: Risk Reduction as Assessed by the World AIDS Foundation (WAF) Risk Reduction Scale
Description: Potentially risky sexual activity and substance use and abuse will be measured using the World AIDS Foundation (WAF) survey Risk Reduction Scale, developed and used with adolescents in South Africa. This measure was adapted for use in Zambia. Score range 8-16. Higher scores indicate feeling more empowered to perform risk reduction intentions, higher scores indicate a better outcome.
Time Frame: Baseline and follow-up within one month of treatment completion. For controls follow up was done 4 months post baseline.
Population: Only participants with complete data were included in this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Wait List Control Group | Intervention Group
Number analyzed (Participants) | 10 | 4
score on a scale
  Baseline | 0.7 (0.4) | 0.9 (0.1)
  Post Assessment | 0.8 (0.4) | 0.2 (0.2)

3. Secondary Outcome: Child Behavior Checklist (CBCL) Score
Description: The CBCL consists of eight empirically-based syndrome subscales. The range of subscale scores (summed) are: Aggressive Behavior (0-36), Anxious/Depressed (0-26), Attention Problems (0-20), Rule-Breaking Behavior (0-34), Somatic Complaints (0-22), Social Problems (0-22), Thought Problems (0-30), and Withdrawn/Depressed (0-16). Score range 0-206. The higher score suggests the more severe symptoms.
Time Frame: Baseline and follow-up within one month of treatment completion. For controls follow up was done 4 months post baseline.
Population: Only participants with complete data were included in this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Wait List Control Group | Intervention Group
Number analyzed (Participants) | 5 | 8
score on a scale
  Baseline | 36.8 (13.0) | 77.8 (48.7)
  Post Assessment | 2.4 (5.4) | 15.8 (14.6)

ADVERSE EVENTS:
Arm/Group | Wait List Control Group | Intervention Group
Serious Adverse Events (participants affected / at risk) | 0/126 | 0/131
Other Adverse Events (participants affected / at risk) | 0/126 | 0/131

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes